CLINICAL TRIAL: NCT01991054
Title: A Prospective, Double Blind, Randomized, Phase 4, Clinical Trial of The Effects of Vitamin D Supplementation on Patients With Type 2 Diabetes and Vitamin D Deficiency
Brief Title: The Effects of Vitamin D Supplementation on Patients With Type 2 Diabetes and Vitamin D Deficiency
Acronym: VDD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, avraham ishay, endocronologist, HaEmek Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HGA1C vs D
Record Dates: First submitted 2013-11-07; First posted 2013-11-25 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2016-09

CONDITIONS: Diabetes Mellitus; Vitamin D Deficiency
Keywords: Diabetes mellitus; HgA1C; 25(OH) vitamin D; HgA1C levels above 7.5%
MeSH Terms: conditions — Diabetes Mellitus; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- vitamin D3 supplementation (Experimental): The study group participants will receive vitamin D3 supplementation (120,000 I.U per month)for 6 months
  Interventions: Dietary Supplement: vitamin D3
- placebo group (Placebo Comparator): placebo group, 15 ml per month for 6 months
  Interventions: Dietary Supplement: vitamin D3

INTERVENTIONS:
Dietary Supplement: vitamin D3
  Other Names: Cholecalciferol

SUMMARY:
Vitamin D plays a key role in keeping normal mineral balance and maintaining bone health. There is accumulating evidence linking deficient vitamin D status with both type 1 and type 2 diabetes.

The purpose of this study is to evaluate the effect of high dose vitamin D supplementation (120000 units per month)for 6 months on glucose homeostasis and glycemic control,in vitamin D deficient patients with non-optimally controlled type 2 diabetes mellitus.

DETAILED DESCRIPTION:
This is a randomized, double blind, parallel group, clinical trial for 6 months duration.

The study group participants will receive vitamin D supplementation (120,000 IU per month) versus the placebo group for 6 months. glycemic control indexes will be measured in T2DM diagnosed study subjects.

Patient will be randomized 1:1 to one of two treatment groups. Vitamin D group vs placebo group.

Randomization kits will include either vitamin D or vitamin D placebo. Blood screens will be taken prior, after 3 months from randomization and after 6 months from randomization. Anthropometric measurements will be drawn as well, at the same time points.

Determination of sample size In order to find a 0.5 mean difference in HgA1C between the two treatment arms (standard deviation 1.2) a 184 sample size will be required to achieve 80% power, 5% alpha (two sided test).

ADMINISTRATIVE AND LEGAL OBLIGATIONS:

Individual patient's medical information obtained as result of this study is considered confidential and disclosure to third parties.

The investigator should maintain a list of appropriately qualified people to whom trail duties are delegated.

Source and study documents will be locked under the supervision of the PI- principle investigator for 15 years.

Study documentations and storage The investigator should maintain a list of appropriately qualified people to whom trail duties are delegated.

All persons authorized to make entries and/or correction on CRF will be included on the investigators team list delegation log.

Study printout and electronic CRF's, ICF's and other study documents will be stored in the at Haemek medical center under the supervision of the PI. All identifying details will be completely erased.

The investigator and staff are responsible for maintaining a comprehensive and centralized filing system of all study- related documentation, suitable for inspection at any time.

ELIGIBILITY:
Inclusion Criteria:

* Written inform consent must be obtained from the patient before any assessment is performed.
* Male or female patient, 18 years or older.
* Diabetes mellitus patients.
* HgA1C levels on randomization above 7.5% in the last 6 months.
* Low 25(OH) vitamin D levels : under 50nmol/l

Exclusion Criteria:

* Patient who are unable consume food orally.
* Life expectancy under 7 month.
* Unable to sign inform consent.
* Patient unwilling or unable to comply with study procedure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Change in Hba1c (%) in study groups | 2 years
  We assume that the treatment with vitamin D will improve diabetes control, as assessed by Hba1c . The expected reduction in Hba1c levels will be 0.5%.

SECONDARY OUTCOMES:
Lipid profile | 2 years
  Total cholesterol, LDL cholesterol , HDL cholesterol, non HDL cholesterol, Triglycerides
C-reactive protein | 2 years
Body Weight | 2 years
Blood Pressure | 2 years
serum calcium | 2 years
serum phosphore | 2 years
serum PTH | 2 years
serum creatinine | 2 years
serum albumin | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: avraham ishay, M.D, Principal Investigator — haemek medical center
Locations (1):
- Haemek medical center, endocrone clinic, Afula, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holick MF. Vitamin D deficiency. N Engl J Med. 2007 Jul 19;357(3):266-81. doi: 10.1056/NEJMra070553. No abstract available. PMID 17634462
- [Background] Bikle D. Nonclassic actions of vitamin D. J Clin Endocrinol Metab. 2009 Jan;94(1):26-34. doi: 10.1210/jc.2008-1454. Epub 2008 Oct 14. PMID 18854395
- [Background] Maalouf NM. The noncalciotropic actions of vitamin D: recent clinical developments. Curr Opin Nephrol Hypertens. 2008 Jul;17(4):408-15. doi: 10.1097/MNH.0b013e3283040c99. PMID 18660678
- [Background] Toubi E, Shoenfeld Y. The role of vitamin D in regulating immune responses. Isr Med Assoc J. 2010 Mar;12(3):174-5. No abstract available. PMID 20684184
- [Background] Peelen E, Knippenberg S, Muris AH, Thewissen M, Smolders J, Tervaert JW, Hupperts R, Damoiseaux J. Effects of vitamin D on the peripheral adaptive immune system: a review. Autoimmun Rev. 2011 Oct;10(12):733-43. doi: 10.1016/j.autrev.2011.05.002. Epub 2011 May 18. PMID 21621002
- [Background] Girgis CM, Clifton-Bligh RJ, Hamrick MW, Holick MF, Gunton JE. The roles of vitamin D in skeletal muscle: form, function, and metabolism. Endocr Rev. 2013 Feb;34(1):33-83. doi: 10.1210/er.2012-1012. Epub 2012 Nov 20. PMID 23169676
- [Background] Wang L, Song Y, Manson JE, Pilz S, Marz W, Michaelsson K, Lundqvist A, Jassal SK, Barrett-Connor E, Zhang C, Eaton CB, May HT, Anderson JL, Sesso HD. Circulating 25-hydroxy-vitamin D and risk of cardiovascular disease: a meta-analysis of prospective studies. Circ Cardiovasc Qual Outcomes. 2012 Nov;5(6):819-29. doi: 10.1161/CIRCOUTCOMES.112.967604. Epub 2012 Nov 13. PMID 23149428
- [Background] Binkley N, Ramamurthy R, Krueger D. Low vitamin D status: definition, prevalence, consequences, and correction. Endocrinol Metab Clin North Am. 2010 Jun;39(2):287-301, table of contents. doi: 10.1016/j.ecl.2010.02.008. PMID 20511052
- [Background] Mithal A, Wahl DA, Bonjour JP, Burckhardt P, Dawson-Hughes B, Eisman JA, El-Hajj Fuleihan G, Josse RG, Lips P, Morales-Torres J; IOF Committee of Scientific Advisors (CSA) Nutrition Working Group. Global vitamin D status and determinants of hypovitaminosis D. Osteoporos Int. 2009 Nov;20(11):1807-20. doi: 10.1007/s00198-009-0954-6. Epub 2009 Jun 19. PMID 19543765
- [Background] Stumvoll M, Goldstein BJ, van Haeften TW. Type 2 diabetes: principles of pathogenesis and therapy. Lancet. 2005 Apr 9-15;365(9467):1333-46. doi: 10.1016/S0140-6736(05)61032-X. PMID 15823385
- [Background] Shaw JE, Sicree RA, Zimmet PZ. Global estimates of the prevalence of diabetes for 2010 and 2030. Diabetes Res Clin Pract. 2010 Jan;87(1):4-14. doi: 10.1016/j.diabres.2009.10.007. Epub 2009 Nov 6. PMID 19896746
- [Background] Takiishi T, Gysemans C, Bouillon R, Mathieu C. Vitamin D and diabetes. Rheum Dis Clin North Am. 2012 Feb;38(1):179-206. doi: 10.1016/j.rdc.2012.03.015. Epub 2012 Apr 12. PMID 22525851
- [Background] Cade C, Norman AW. Vitamin D3 improves impaired glucose tolerance and insulin secretion in the vitamin D-deficient rat in vivo. Endocrinology. 1986 Jul;119(1):84-90. doi: 10.1210/endo-119-1-84. PMID 3013599
- [Background] Norman AW, Frankel JB, Heldt AM, Grodsky GM. Vitamin D deficiency inhibits pancreatic secretion of insulin. Science. 1980 Aug 15;209(4458):823-5. doi: 10.1126/science.6250216.
- [Background] Norman AW. Minireview: vitamin D receptor: new assignments for an already busy receptor. Endocrinology. 2006 Dec;147(12):5542-8. doi: 10.1210/en.2006-0946. Epub 2006 Aug 31. PMID 16946007
- [Background] Maestro B, Davila N, Carranza MC, Calle C. Identification of a Vitamin D response element in the human insulin receptor gene promoter. J Steroid Biochem Mol Biol. 2003 Feb;84(2-3):223-30. doi: 10.1016/s0960-0760(03)00032-3. PMID 12711007
- [Background] Maestro B, Molero S, Bajo S, Davila N, Calle C. Transcriptional activation of the human insulin receptor gene by 1,25-dihydroxyvitamin D(3). Cell Biochem Funct. 2002 Sep;20(3):227-32. doi: 10.1002/cbf.951. PMID 12125099
- [Background] Dunlop TW, Vaisanen S, Frank C, Molnar F, Sinkkonen L, Carlberg C. The human peroxisome proliferator-activated receptor delta gene is a primary target of 1alpha,25-dihydroxyvitamin D3 and its nuclear receptor. J Mol Biol. 2005 Jun 3;349(2):248-60. doi: 10.1016/j.jmb.2005.03.060. Epub 2005 Apr 7. PMID 15890193
- [Background] Maestro B, Campion J, Davila N, Calle C. Stimulation by 1,25-dihydroxyvitamin D3 of insulin receptor expression and insulin responsiveness for glucose transport in U-937 human promonocytic cells. Endocr J. 2000 Aug;47(4):383-91. doi: 10.1507/endocrj.47.383. PMID 11075718
- [Background] Pittas AG, Lau J, Hu FB, Dawson-Hughes B. The role of vitamin D and calcium in type 2 diabetes. A systematic review and meta-analysis. J Clin Endocrinol Metab. 2007 Jun;92(6):2017-29. doi: 10.1210/jc.2007-0298. Epub 2007 Mar 27. PMID 17389701
- [Background] Scragg R, Sowers M, Bell C; Third National Health and Nutrition Examination Survey. Serum 25-hydroxyvitamin D, diabetes, and ethnicity in the Third National Health and Nutrition Examination Survey. Diabetes Care. 2004 Dec;27(12):2813-8. doi: 10.2337/diacare.27.12.2813. PMID 15562190
- [Background] Muscogiuri G, Sorice GP, Ajjan R, Mezza T, Pilz S, Prioletta A, Scragg R, Volpe SL, Witham MD, Giaccari A. Can vitamin D deficiency cause diabetes and cardiovascular diseases? Present evidence and future perspectives. Nutr Metab Cardiovasc Dis. 2012 Feb;22(2):81-7. doi: 10.1016/j.numecd.2011.11.001. Epub 2012 Jan 21. PMID 22265795
- [Background] Oosterwerff MM, Eekhoff EM, Heymans MW, Lips P, van Schoor NM. Serum 25-hydroxyvitamin D levels and the metabolic syndrome in older persons: a population-based study. Clin Endocrinol (Oxf). 2011 Nov;75(5):608-13. doi: 10.1111/j.1365-2265.2011.04110.x. PMID 21595731
- [Background] Husemoen LL, Skaaby T, Thuesen BH, Jorgensen T, Fenger RV, Linneberg A. Serum 25(OH)D and incident type 2 diabetes: a cohort study. Eur J Clin Nutr. 2012 Dec;66(12):1309-14. doi: 10.1038/ejcn.2012.134. Epub 2012 Oct 3. PMID 23031851
- [Background] Forouhi NG, Luan J, Cooper A, Boucher BJ, Wareham NJ. Baseline serum 25-hydroxy vitamin d is predictive of future glycemic status and insulin resistance: the Medical Research Council Ely Prospective Study 1990-2000. Diabetes. 2008 Oct;57(10):2619-25. doi: 10.2337/db08-0593. Epub 2008 Jun 30. PMID 18591391
- [Background] Knekt P, Laaksonen M, Mattila C, Harkanen T, Marniemi J, Heliovaara M, Rissanen H, Montonen J, Reunanen A. Serum vitamin D and subsequent occurrence of type 2 diabetes. Epidemiology. 2008 Sep;19(5):666-71. doi: 10.1097/EDE.0b013e318176b8ad. PMID 18496468
- [Background] Robinson JG, Manson JE, Larson J, Liu S, Song Y, Howard BV, Phillips L, Shikany JM, Allison M, Curb JD, Johnson KC, Watts N. Lack of association between 25(OH)D levels and incident type 2 diabetes in older women. Diabetes Care. 2011 Mar;34(3):628-34. doi: 10.2337/dc10-1632. Epub 2011 Feb 2. PMID 21289227
- [Background] Boucher BJ, Mannan N, Noonan K, Hales CN, Evans SJ. Glucose intolerance and impairment of insulin secretion in relation to vitamin D deficiency in east London Asians. Diabetologia. 1995 Oct;38(10):1239-45. doi: 10.1007/BF00422375. PMID 8690178
- [Background] Borissova AM, Tankova T, Kirilov G, Dakovska L, Kovacheva R. The effect of vitamin D3 on insulin secretion and peripheral insulin sensitivity in type 2 diabetic patients. Int J Clin Pract. 2003 May;57(4):258-61. PMID 12800453
- [Background] Orwoll E, Riddle M, Prince M. Effects of vitamin D on insulin and glucagon secretion in non-insulin-dependent diabetes mellitus. Am J Clin Nutr. 1994 May;59(5):1083-7. doi: 10.1093/ajcn/59.5.1083. PMID 8172095
- [Background] Major GC, Alarie F, Dore J, Phouttama S, Tremblay A. Supplementation with calcium + vitamin D enhances the beneficial effect of weight loss on plasma lipid and lipoprotein concentrations. Am J Clin Nutr. 2007 Jan;85(1):54-9. doi: 10.1093/ajcn/85.1.54. PMID 17209177
- [Background] Fliser D, Stefanski A, Franek E, Fode P, Gudarzi A, Ritz E. No effect of calcitriol on insulin-mediated glucose uptake in healthy subjects. Eur J Clin Invest. 1997 Jul;27(7):629-33. doi: 10.1046/j.1365-2362.1997.1520699.x. PMID 9263752
- [Background] Grimnes G, Joakimsen R, Figenschau Y, Torjesen PA, Almas B, Jorde R. The effect of high-dose vitamin D on bone mineral density and bone turnover markers in postmenopausal women with low bone mass--a randomized controlled 1-year trial. Osteoporos Int. 2012 Jan;23(1):201-11. doi: 10.1007/s00198-011-1752-5. Epub 2011 Sep 10. PMID 21909730
- [Background] Pittas AG, Harris SS, Stark PC, Dawson-Hughes B. The effects of calcium and vitamin D supplementation on blood glucose and markers of inflammation in nondiabetic adults. Diabetes Care. 2007 Apr;30(4):980-6. doi: 10.2337/dc06-1994. Epub 2007 Feb 2. PMID 17277040
- [Background] Nagpal J, Pande JN, Bhartia A. A double-blind, randomized, placebo-controlled trial of the short-term effect of vitamin D3 supplementation on insulin sensitivity in apparently healthy, middle-aged, centrally obese men. Diabet Med. 2009 Jan;26(1):19-27. doi: 10.1111/j.1464-5491.2008.02636.x. PMID 19125756
- [Background] George PS, Pearson ER, Witham MD. Effect of vitamin D supplementation on glycaemic control and insulin resistance: a systematic review and meta-analysis. Diabet Med. 2012 Aug;29(8):e142-50. doi: 10.1111/j.1464-5491.2012.03672.x. PMID 22486204
- [Background] Bischoff-Ferrari HA, Giovannucci E, Willett WC, Dietrich T, Dawson-Hughes B. Estimation of optimal serum concentrations of 25-hydroxyvitamin D for multiple health outcomes. Am J Clin Nutr. 2006 Jul;84(1):18-28. doi: 10.1093/ajcn/84.1.18. PMID 16825677
- [Background] Aloia JF, Patel M, Dimaano R, Li-Ng M, Talwar SA, Mikhail M, Pollack S, Yeh JK. Vitamin D intake to attain a desired serum 25-hydroxyvitamin D concentration. Am J Clin Nutr. 2008 Jun;87(6):1952-8. doi: 10.1093/ajcn/87.6.1952. PMID 18541590
- [Background] Holick MF, Binkley NC, Bischoff-Ferrari HA, Gordon CM, Hanley DA, Heaney RP, Murad MH, Weaver CM; Endocrine Society. Evaluation, treatment, and prevention of vitamin D deficiency: an Endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2011 Jul;96(7):1911-30. doi: 10.1210/jc.2011-0385. Epub 2011 Jun 6. PMID 21646368
- See also: 41. "Vitamin D and Calcium: Updated Dietary Reference Intakes". Nutrition and Healthy Eating. Health Canada. Retrieved 2012-06-13. — http://www.hc-sc.gc.ca/fn-an/nutrition/vitamin/vita-d-eng.php
- See also: 42. U.S. Food and Drug Administration: Guidance for Industry: A Food labeling Guide. — http://www.fda.gov.